CLINICAL TRIAL: NCT06460649
Title: Combined Effects Of Progressive Relaxation Techniques Along With Benson Relaxation Techniques on Stress Fatigue and Quality of Life on Postpartum Females
Brief Title: Combined Effects Of Progressive Relaxation Techniques Along With Benson Relaxation Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0586
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Postpartum Disorder
Keywords: Fatigue; Postpartum relaxation techniques; Postpartum period; Postpartum women; Quality of life; Stress
MeSH Terms: conditions — Puerperal Disorders; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation techniques+Benson relaxation techniques (Experimental): Participants in group A will receive progressive relaxation techniques along benson relaxation sessions will be conducted 3 times a week for 12 weeks . Total number of sessions will be 3
  Interventions: Other: Progressive relaxation techniques; Other: Benson relaxation techniques
- Progressive relaxation techniques (Active Comparator): Participants in group B will receive progressive relaxation techniques only. Sessions will be conducted 3 times a week for 12 weeks.36 sessions over all
  Interventions: Other: Progressive relaxation techniques

INTERVENTIONS:
Other: Progressive relaxation techniques — Participants received Progressive muscle relaxation along with Benson relaxing 3 times a week for 12 weeks. 36 sessions overall
Other: Benson relaxation techniques — Participants received Benson relaxation techniques 3 times a week for 12 weeks. 36 sessions overall.
  Arms: Progressive relaxation techniques+Benson relaxation techniques

SUMMARY:
The postpartum (or postnatal) period begins after childbirth and is typically considered to last for six weeks. Stress is considered a response to any stressor within external or internal milieu, to stay in an adaptive mode using functional or dysfunctional coping skills. It initiates an alterable mode that ultimately becomes a prolonged adaptive struggle The study will be a randomized controlled trial and will be conducted in Jinnah hospital, Lahore. This study will be completed in a time duration of 8 months after the approval of synopsis. Nonprobability convenience sampling technique will be used, and participants will be recruited in study after randomization. The subjects will be divided into two groups and group A will receive progressive relaxation technique along with Benson relaxing technique. and group B will receive progressive relaxation technique and deep breathing exercises will be used as a baseline treatment. The tools that will be used for pre and post treatment assessment are Postpartum fatigue scale (PFS), Perceived Stress Scale (PSS_10), WHOQOL-BREF Scale. The data will be assessed after 12 weeks. After data collection data will be analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
The postpartum (or postnatal) period begins after childbirth and is typically considered to last for six weeks. Postpartum period can be a challenging time for many women, as they often experience increased stress levels, fatigue, and a change in their overall quality of life. Stress is considered a response to any stressor within external or internal milieu, to stay in an adaptive mode using functional or dysfunctional coping skills. It initiates an alterable mode that ultimately becomes a prolonged adaptive struggle when an individual cannot find the right coping skills, which may then become a long term dysfunctional state, hence a chronic psychiatric condition.

The study will be a randomized controlled trial and will be conducted in Jinnah hospital, Lahore. This study will be completed in time duration of 5_6 months after the approval of synopsis. Non probability convenience sampling technique will be used and participants will be recruited in study after randomization. The subjects will be divided into two groups and the group A will receive progressive relaxation technique along with Benson relaxing technique. and group B will receive progressive relaxation technique and deep breathing exercises will be used as a baseline treatment. The tools that will be used for pre and post treatment assessment are Postpartum fatigue scale(PFS), Perceived Stress Scale (PSS_10), WHOQOL-BREF Scale. The data will be assessed after 5 days 45min per treatment session. After data collection data will be analyzed by using SPSS version 25.

Key words: Fatigue, progressive Relaxation technique, Postpartum period, Postpartum women, Quality of life, Stress

ELIGIBILITY:
Inclusion Criteria:

* • Parity of women must not more than 3 times

  * Start from 2nd week of postpartum female
  * Women with aged group of 20- 40 were included in study.(24)
  * Women who had Vaginal or c section delivery were included in study.
  * Women with no postnatal complications were included in study

Exclusion Criteria:

* • Women with Diabetes Militias were excluded

  * Women with Breast cancer were excluded
  * Ovarian cancer were excluded
  * Patient with dementia, delusional disorder were excluded
  * Women who use Alcohol or substance abuse were excluded
  * Women who had a history of psychiatric disorders were excluded
  * Severed obesity ( BMI more than 40)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female (postpartum)
Enrollment: 54 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Postpartum fatigue scale | 12 weeks
  Postpartum fatigue scale four-point scale to respond to the PFS questionnaire, which included-physical stress, mental stress, sleep deprivation, exploratory factor analysis, it was determined that PAFS consisted of 13 items, 6 items in the "Physical Fatigue" subdimension, 4 items in the "Emotional" subdimension, and 3 items in the "Cognitive" subdimension. The three-factor scale structure supported confirmatory factor analysis. On the total scale, Cronbach's α was found to be 0.91.(24)
Perceived stress scale | 12 weeks
  The Perceived Stress Scale (PSS) is a classic stress assessment instrument. The tool, while originally developed in 1983,. The questions in this scale ask about your feelings and thoughts during the last month.. The best approach is to answer fairly quickly. That is, don't try to count up the number of times you felt a particular way; rather indicate the alternative that seems like a reasonable estimate Figuring Your PSS Score You can determine your PSS score by following these directions: • First, reverse your scores for questions 4, 5, 7, and 8.
  On these 4 questions, change the scores like this: 0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0.
WHOQOL-BREF Scale | 12 weeks
  The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) is an abbreviated, 26-item version of the 100-item WHOQOL-100 quality of life measure. The
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items);. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale . The physical health domain includes items on mobility, daily activities, functional capacity, energy, pain, and sleep. the 8-item the reliability of the WHOQOL-5 was below the acceptable threshold (PSI = 0.66). Reliability of the EUROHIS-QOL-8 was satisfactory (PSI = 0.79)(24)

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.phill, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No